CLINICAL TRIAL: NCT02305576
Title: Effect of Perioperative Factors on the Analgesia Nociception Index
Acronym: ANIFACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 13-181
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Analgesia Nociception Index (ANI) is a new unitless marker derived from Heart Rate Variability spectral analysis, ranging between 0 and 100 and expressing the parasympathetic tone. The ANI is proposed as surrogate marker for the analgesia nociception balance. However, many perioperative factors such as medications, position, maneuvers may influence the ANI values and may lead to misinterpretation. Moreover the ability of the ANI to guide opioid dosing has never been tested. Therefore, the aim of our study is to collect in a database all the perioperative factors and to study their influence on the ANI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled surgery

Exclusion Criteria:

* Non sinusal rhythm
* Pace maker or defibrillator holders
* Pregnancy or feeding
* American Society of Anesthesiology physical status 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patietns undergoing planned surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation of the ANI index | Before and 2 minutes afer the factor occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Georges Daccache, M.D, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, Calvados, France